CLINICAL TRIAL: NCT03416348
Title: Hyperhidrosis of the Residual Limb in Patients With Amputations: Developing a Treatment Approach, Aims 1 and Aim 2
Brief Title: Hyperhidrosis, Developing a Treatment Approach Aims 1 & 2
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Responsible Party: Principal Investigator, Colby Hansen, Principle Investigator, University of Utah
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: OP150030 (Aim 1&2); OP150030 (Other Grant/Funding Number: DOD)
Record Dates: First submitted 2017-12-19; First posted 2018-01-31 (Actual); Last update posted 2022-10-17 (Actual); Status verified 2022-10

CONDITIONS: Hyperhidrosis
Keywords: amputation; amputations; sweating; residual limb; service members; civilians
MeSH Terms: conditions — Hyperhidrosis | interventions — Aluminum Chloride; Deodorants; Ethanol

STUDY DESIGN:
Intervention Model Description: For the two aims of the study, subjects will be recruited from the amputee clinics held at the Salt Lake VA Medical Center or the University of Utah. Combined, these clinics serve approximately 500 patients and see approximately 75 new patients each year. Based on the investigators work, which showed 66% of patients with HDSS scores of 2 or greater, we will have a potential pool of up to 330 eligible patients for the studies that follow. We expect to enroll approximate equal numbers from both sites for each of the aims of this study.
Who Masked: Participant, Investigator
Masking Description: For Aim 1 there will be no masking. Aim 2, recruitment methods will be by convenience sampling. Subjects in Aim 1 reporting an HDSS of 2 or greater and additional subjects as needed from the U of U or VA clinics with HDSS of 2 or greater will be invited to participate in this crossover study. Subjects will be randomized equally to two sequence arms by a random number generator. The first arm will receive in sequential order every 3 weeks: Aluminum Chloride, a placebo of ethyl alcohol base, Aluminum Chloride, and placebo. The second arm will receive in sequential order every 3 weeks: placebo, Aluminum Chloride, placebo, and Aluminum Chloride. Each condition will last for 3 weeks, which will allow enough time for the Aluminum Chloride and placebo to demonstrate their respective effects. The first week of each period will also serve as a sufficient washout for the previous period. The total trial length, then, will be 12 weeks.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo Comparator AIM 1 (Placebo Comparator): Aim 1: Demonstration of a strong association of the Sweating Intensity Visual Scale (SIVS) score with the HDSS would provide validation for use of the SIVS in interpreting the iodine-starch test and would establish the value of the iodine-starch test in clinical practice guidelines for diagnosing hyperhidrosis in amputees, just as it is in dermatology practice.
  Interventions: Drug: Aluminum Chloride 20% (deodorant); Drug: Alcohol
- Aluminum Chloride vs Placebo in Amputees (Active Comparator): Aim 2: The investigators will have completed the first clinical trial of Aluminum Chloride for residual limb hyperhidrosis. The investigators will then have a solid foundation of data that demonstrates the rates of adverse effects such as skin irritation, and rates and magnitudes of improvement in subjective and objective measures of sweating.
  Interventions: Drug: Aluminum Chloride 20% (deodorant); Drug: Alcohol

INTERVENTIONS:
Drug: Aluminum Chloride 20% (deodorant) — Aluminum Chloride (deodorant)
  Other Names: Drysol, XeracAC
Drug: Alcohol — Placebo
  Other Names: Ethyl Alcohol

SUMMARY:
The objective is to establish an evidence base for a hyperhidrosis treatment algorithm in amputees. This project will address a problem that has troubled Service members, Veterans, and civilians with amputations for decades, impacting satisfaction with prosthetic use, residual limb skin health, and negatively affecting quality of life. Prior research in this area has been limited and insufficient. The Investigators are confident that improving the evaluation and treatment of residual limb hyperhidrosis will reduce the secondary health consequences of amputation and will lead to improved quality of life. This will be accomplish by completing the following specific aims.

Aim 1: Test the validity of the Minor iodine-starch test in amputees. Hypothesis: The iodine-starch test is a valid diagnostic tool of hyperhidrosis and can be useful for the identification of focal areas of sweating on a residual limb Aim 2: Test the effectiveness of a prescription strength topical antiperspirant (Aluminum Chloride 20%) on hyperhidrosis of the residual limb.

Hypothesis: Aluminum Chloride will be more effective at controlling sweating than placebo

DETAILED DESCRIPTION:
One objective of the Prosthetic Outcomes Research Award (PORA) is to improve the understanding of secondary health effects on Service members and Veterans who have undergone limb amputation and to advance the adoption and implementation of evidence-based interventions. The investigators will address the important secondary health problem of excessive residual limb sweating (hyperhidrosis) in amputees.

Successful use of a prosthesis requires a stable interface between the residual limb and the prosthetic socket. Maintaining healthy skin, therefore, is paramount. However, the closed environment necessary to provide this stable interface also creates an environment that may lead to a multitude of skin problems. Amputees regularly deal with skin problems such as sweating, eczematous itching and redness, infections, and mechanical problems such as blisters and open wounds. Hyperhidrosis is the single most reported problem. Hyperhidrosis is reported in up to 70% of amputee and is associated with reduced quality of life, reduced prosthetic fit and function, decreased satisfaction with their prosthesis and skin irritation. The investigators own published findings reveal that 66% of prosthetic users (both veteran and civilian) experienced residual limb sweating that interfered with activities of daily living. Sweating was rated as most bothersome in warm weather or with vigorous activity, and the efficacy of treatment strategies was generally reported to be poor.

Despite the frequency and impact of hyperhidrosis in amputees, there is a lack of evidence based guidelines for evaluating and treating this problem. A number of knowledge gaps exist, including no clear standard for assessing the burden of sweating in amputees, and no evidence base from which to inform treatment decisions for either simple or more elaborate interventions.

There is no universally accepted standard for assessing the burden and precise location of sweating in amputee patients. Among the several subjective scales of hyperhidrosis severity in the dermatology literature, the most commonly used and rigorously validated one is the Hyperhidrosis Disease Severity Scale (HDSS). The HDSS provides a qualitative measure for the severity of the patient's condition based on the extent to which hyperhidrosis affects daily activities. The HDSS is simple to administer and scored as follows:

Hyperhidrosis Disease Severity Scale

Condition:

Score

1. My sweating is never noticeable and never interferes with my daily activities
2. My sweating is tolerable but sometimes interferes with my daily activities
3. My sweating is barely tolerable and frequently interferes with my daily activities
4. My sweating is intolerable and always interferes with my daily activities

In the general hyperhidrosis patient population (non-amputee), the HDSS exhibits moderate to strong correlations with other quality of life and disease impact metrics, as well as with gravimetric sweat production. A 1 point improvement on the HDSS correlates with a 50% reduction in sweat production, while a 2 point improvement correlates with an 80% reduction in sweat production. The investigators survey data shows the HDSS correlates well with amputees' perception of the impact of sweating on their prosthesis fit and function, and is therefore a valid outcome measure in the amputee population.

While the HDSS gives a global, patient-reported outcome of the significance of hyperhidrosis in the patient's life, it does not inform the treating clinician on the precise location of the problem. Dermatologists treating hyperhidrosis of other regions (i.e. axillary, palmar, plantar) use the Minor iodine-starch test to identify the area of hyperhidrosis in order to guide subsequent treatments. This test consists of an application of iodine, which is allowed to dry and then dusted with cornstarch. Sweat will react with the iodine and starch and produce a black/purple color. While this test is primarily used to identify the areas of hyperhidrosis, a grading scale has been proposed for test interpretation and monitoring response to treatments. There is scant literature describing the iodine-starch test in amputees and the investigators early experience suggests that it is insufficient to simply apply iodine and starch on a residual limb without then donning the patient's prosthesis. It appears necessary to recreate the environment that produces the excessive sweating by donning the prosthesis and ambulating. It is not known, however, what method is safe and effective, without causing harm to the patient's skin and/or prosthetic materials.

As part of the scope of the research proposed herein, the investigators have done pilot work with 9 subjects and 11 amputation sites, utilizing the iodine-starch test under a variety of conditions to assess which method is most feasible to allow the patient to use their prosthesis in the test. Preliminary results suggest that plastic wrap is adequate to protect the prosthesis from significant iodine stain and does not cause new skin irritation, but is more often viewed as uncomfortable. It also appears to induce a very rapid and diffuse pattern sweating, raising concern for creating too much of a false positive effect. A prosthetic sheath appears to protect the liner from dense stain, though some light iodine stain has been observed to seep onto the liner in some cases. This method, though, is generally viewed as comfortable to the patient, does not cause new skin irritation, and does produce a positive test after 10 - 15 minutes of walking in focal areas more consistent with the patient's described experience with sweat and sweat location.

The investigators believe that applying the iodine-starch combination, donning a prosthetic sheath, the patient's own prosthesis, followed by a period of ambulation is the best method for future studies.

Beyond the assessment of hyperhidrosis, treatment guidelines for this problem have not been rigorously applied to amputees. In the dermatology literature, guidelines recommend using a topical antiperspirant such as Aluminum Chloride (AlCl) as first line treatment. For axillary hyperhidrosis, treatment success with AlCl (defined as a post treatment HDSS score of 1, has varied from 33% to 72% in clinical trials). However, in the amputee population, there are no published clinical trials describing the effectiveness or tolerability of a topical treatment, and if it is ineffective or intolerable, when to consider another option such as botulinum toxin injections, which are generally considered as second line treatment. The investigators found through a survey that 50% of respondents had tried either an over the counter or prescription strength antiperspirant. Of those respondents having tried such an agent, nearly 50% reported them to have no efficacy, and only about 20% reported them to be completely or mostly effective. Clearly this data has limitations, due to subject recall bias, and is not the product of an intervention study. It does, however, illustrate that a majority of amputees may not have satisfactory options to treat this problem.

There have been a few case reports and/or case series reporting the use of botulinum toxin to treat this problem in amputees. While these preliminary reports suggest that botulinum toxin is an effective treatment option, they are limited by the fact that the intervention was tried on such a small number of patients. Kern et al used botulinum toxin type B (BTX-B) in 9 patients while Charrow et al. used botulinum toxin type A (BTX-A) in 8 patients. Both reported good effectiveness in treating hyperhidrosis but neither utilized a validated method to determine effectiveness, nor did the subjects fail a topical treatment prior to botulinum toxin treatment.

Further, there is no published literature describing the best way to localize botulinum toxin application for amputee hyperhidrosis. In considering the feasibility of widespread adoption of botulinum toxin as a treatment for amputee hyperhidrosis, one of the biggest barriers could be the large surface area involved that needs to be treated.

Dermatologists use the iodine-starch test to identify the hyperhidrotric area that will be targeted with the botulinum toxin injection. For palmar, axillary, and plantar hyperhidrosis, it is recommended that every patient be assessed with this method. A single case study has reported the successful use of the iodine-starch test to help identify hyperhidrotic areas on a residual limb. However, it has not been well studied to know if the iodine-starch test can be utilized in amputees to identify potential sites for injection, or even if the pattern of sweating can be demonstrated to be a focal, not a global, problem. If the iodine-starch test can be used successfully in amputees, it could help direct botulinum toxin injections to a focused area, rather than an entire residual limb. This could have significant impact on the overall tolerability of the procedure and the willingness of both patients and providers to implement it in usual clinical care.

ELIGIBILITY:
Aim 1 and Aim 2

Inclusion Criteria:

* Provision of signed and dated informed consent form (ICF)
* Stated willingness to comply with all study procedures and availability for the duration of the study
* Male or female, age 18 or older
* Have a prosthetic device
* In good general health as evidenced by medical history
* If subject is currently using aluminum chloride participant must be discontinued for at least one week prior to participation in the study.

Exclusion Criteria:

* Open sores or wounds on the residual limb
* Known sensitivity or allergy to iodine
* Known sensitivity to antiperspirant, aluminum chloride hexahydrate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2018-05-08 (Actual); Primary Completion 2022-01-15 (Actual); Study Completion 2022-02-14 (Actual)

PRIMARY OUTCOMES:
Hyperhidrosis Disease Severity Scale (HDSS) | 1 day
  The outcome measure of Aim 1 will be measuring the Hyperhidrosis Disease Severity Scale (HDSS). The HDSS is scored on a number scale of 1-4. Score range from 1 (lowest) demonstrating sweating (hyperhidrosis) is least noticeable and does not interfere with daily activities (least impactful) to 4 (highest) sweating is intolerable and interferes significantly with daily activities. This measurement will be completed in a single site visit.

SECONDARY OUTCOMES:
Hyperhidrosis Disease Severity Scale (HDSS) | 12 weeks
  The outcome measure of Aim 2 will be measuring the Hyperhidrosis Disease Severity Scale (HDSS) in a cross over design at 12 weeks of those participants with an HDSS score of 2 or higher. The HDSS is scored on a number scale of 1-4. Score range from 1 (lowest) demonstrating sweating (hyperhidrosis) is least noticeable and does not interfere with daily activities (least impactful) to 4 (highest) sweating is intolerable and interferes significantly with daily activities.

CONTACTS AND LOCATIONS:
Overall Officials: Colby Hansen, MD, Principal Investigator — University of Utah
Locations (2):
- United States (2):
  - George E. Wahlen Department of Veterans Affairs Medical Center, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No